CLINICAL TRIAL: NCT01319656
Title: Adaptation, Implementation and Evaluation of an Intervention Involving the Integration of Chronic Disease Rehabilitation Services Into Primary Care
Brief Title: Integration of Chronic Disease Rehabilitation Services Into Primary Care
Acronym: PR1MaC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Fortin (Other)
Collaborators: Pfizer (Industry); Fonds de la Recherche en Santé du Québec (Other Government); Ministere de la Sante et des Services Sociaux (Other); Centre de santé et de services sociaux de Chicoutimi (Other); Centre de santé et de services sociaux de Jonquière (Other)
Responsible Party: Sponsor-Investigator, Martin Fortin, Dr, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: FRSQ-24423
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Disease; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Diabetes
Keywords: Chronic diseases; Primary care; Rehabilitation; Chronic Care Model; Patient centered medical home
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Diabetes Mellitus; Chronic Disease | interventions — Palliative Care; Therapeutics; Counseling; Respiratory Therapy; Exercise; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Intervention group(n = 163)
  Interventions: Behavioral: Support, management, educational, counselling, follow-up
- Group B (Active Comparator): Delayed intervention (n = 163)
  Interventions: Behavioral: Support, management, educational, counselling, follow-up
- Group C (No Intervention): No intervention group (n = 163)

INTERVENTIONS:
Behavioral: Support, management, educational, counselling, follow-up — The project offers a range of activities (educational, counselling, follow-up) by several professionals. The varied range of services is spread out over six months and may include individual or group meetings with professionals. Informational documents and follow-up tools are provided to patients based on their condition, to facilitate the acquisition and maintenance of knowledge, self-management, and changes in risk behaviour.
  Other Names: dietetics, respiratory therapy, smoking cessation, physical activity, Stress management, Psychosocial support, Drug compliance
  Arms: Group A; Group B

SUMMARY:
The aim of PR1MaC is to establish a clinical intervention that will adapt and permanently integrate rehabilitation services into primary care settings, which would be the reference point in the health care system for people with Chronic diseases (CD). More specifically, the intervention will aim to: (1) clinically operationalize the mechanisms and tools necessary for delivery of integrated CD services, promoting continuity of care in response to the needs expressed by stakeholders; (2) implement and deploy rehabilitation services adapted to the realities of various clinical primary care settings and develop tools to ensure the sustainability of interventions beyond the rehabilitation period; and (3) support clinical primary care teams in the acquisition and maintenance of evidence-based practices for the targeted CDs.

DETAILED DESCRIPTION:
Since 2001, professionals in the Saguenay-Lac-Saint-Jean (SLSJ) region in Quebec province, Canada, have been mobilized to deal with the challenges of CD management by the introduction of the SLSJ Trajectory of Integrated Rehabilitation Services for CD (Trajectoire des services de réadaptation intégrés pour MC du SLSJ), hereafter referred to as the "Trajectoire." This Trajectoire, deployed across the region, constitutes a solid network of rehabilitation services, due as much to the resources granted to it and its evidence-based approach as to the appreciation that patients and professionals within the regional health system have for it. The changes and new directions that have taken place in recent years suggest it is time to improve this Trajectoire by promoting greater integration with primary care services to improve accessibility, the complementarity of services and better post-rehabilitation continuity. The proposed intervention involves the adaptation and integration of rehabilitation services under the Trajectoire's leadership within primary care settings (FMG or medical clinics), so that collaborative work routines are developed and implemented directly at the main place of contact with health services for people with a CD. The intervention will be implemented at the CSSSs in Chicoutimi and Jonquière. This logic model was developed in collaboration with researchers, clinicians and decision-makers involved in this application and discussed at meetings for the preparation of this application. The model's first component (objective 1) will consist of a consultation with stakeholders (primary care professionals, Trajectoire professionals) by sharing information about the current range of services. In each area, the consultation will include a needs evaluation and a reflection on the Trajectoire's services that can be adapted for targeted clients. As each clinic where an intervention will be deployed has its own mode of operation and clientele characteristics, the clinical intervention will be specifically adapted to these considerations and prepared in collaboration with each clinical setting to ensure a range of services that meets the expressed needs.

The second component (objective 2) will be to implement and deploy a range of concerted interdisciplinary services adapted to the client services and professional resources already in place. Services that do not require specialized equipment or adapted premises (a gym, for example) can be integrated, including educational/teaching services (self-care, support to stop smoking, nutrition, etc.). In medical clinics currently not offering these services, the addition will be net, while in those that already rely on the services of nurse practitioners (FMG), the addition of these services will complement existing services. During this period, various mechanisms and clinical information sharing tools will be implemented jointly by professionals. The third component will be to implement a support mechanism and ongoing evaluation within the clinical setting to ensure harmonious integration. If necessary, training workshops will be provided to implement or maintain evidence-based practices and to plan longer-term follow-up of clientele and continuity of interventions.

The intervention: (a) will be educational in nature, patient-centred and based on the Trajectoire; (b) will last at least three months and involve at least three meetings; (c) may include meetings with small patient groups or the involvement of a close relative of the patient (spouse or primary caregiver); (d) will be carried out based on a referral from the primary care team according to defined criteria; (e) will allow an exchange with the primary care team and will be integrated into the primary care medical records; (f) will provide for a transfer of responsibility to the primary care team to ensure ongoing long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* present at least one of the following conditions: type 2 diabetes, CVD, heart failure, risk factors (smoking, obesity, hyperlipidemia, glucose intolerance, and metabolic syndrome), COPD or asthma.
* have the potential for rehabilitation

Exclusion Criteria:

* serious cognitive problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of effects | T1: Initial evaluation; T2: after three months; T3: one year after T1
  Short term:
  * Self-Efficacy Managing Chronic Disease scale: SEMCD
  * Health Education Impact questionnaire: heiQ
  Medium term:
  * Risk factors
  * Functional health status/quality of life: SF12
  * Psychological well being: K6
  Other:
  * Socio-demographic: SD
  * comorbidity
  * co-intervention (CI)
  Visites:
  * 1:(week:- 2) : Group A and B: DBMA; SD; SF12; K6; SEMCD, heiQ
  * 2a:(week:0) : Group A, (week:12) for Group B: SEMCD, heiQ; CI
  * 2b, 2c: (weeks:4, 8) : Group A: CI
  * 3:(weeks:12) : Group A: SEMCD, heiQ; CI
  * 4:(weeks:52) : Group A: SF12, K6; SEMCD, heiQ; CI

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fortin, MD, M.Sc., Principal Investigator — Université de Sherbrooke
Locations (1):
- CSSS de Chicoutimi, Unité de médecine de famille, Chicoutimi, Quebec, Canada

REFERENCES:
- [Background] Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff (Millwood). 2001 Nov-Dec;20(6):64-78. doi: 10.1377/hlthaff.20.6.64. PMID 11816692
- [Background] Tsai AC, Morton SC, Mangione CM, Keeler EB. A meta-analysis of interventions to improve care for chronic illnesses. Am J Manag Care. 2005 Aug;11(8):478-88. PMID 16095434
- [Background] Dennis SM, Zwar N, Griffiths R, Roland M, Hasan I, Powell Davies G, Harris M. Chronic disease management in primary care: from evidence to policy. Med J Aust. 2008 Apr 21;188(S8):S53-6. doi: 10.5694/j.1326-5377.2008.tb01745.x. PMID 18429737
- [Background] Rothman AA, Wagner EH. Chronic illness management: what is the role of primary care? Ann Intern Med. 2003 Feb 4;138(3):256-61. doi: 10.7326/0003-4819-138-3-200302040-00034. PMID 12558376
- [Background] Chreim S, Williams BE, Janz L, Dastmalchian A. Change agency in a primary health care context: the case of distributed leadership. Health Care Manage Rev. 2010 Apr-Jun;35(2):187-99. doi: 10.1097/HMR.0b013e3181c8b1f8. PMID 20234224
- [Background] Hogg W, Lemelin J, Moroz I, Soto E, Russell G. Improving prevention in primary care: Evaluating the sustainability of outreach facilitation. Can Fam Physician. 2008 May;54(5):712-20. PMID 18474705
- [Background] Clark AM, Hartling L, Vandermeer B, McAlister FA. Meta-analysis: secondary prevention programs for patients with coronary artery disease. Ann Intern Med. 2005 Nov 1;143(9):659-72. doi: 10.7326/0003-4819-143-9-200511010-00010. PMID 16263889
- [Background] Peytremann-Bridevaux I, Staeger P, Bridevaux PO, Ghali WA, Burnand B. Effectiveness of chronic obstructive pulmonary disease-management programs: systematic review and meta-analysis. Am J Med. 2008 May;121(5):433-443.e4. doi: 10.1016/j.amjmed.2008.02.009. PMID 18456040
- [Background] Gibson PG, Powell H, Coughlan J, Wilson AJ, Abramson M, Haywood P, Bauman A, Hensley MJ, Walters EH. Self-management education and regular practitioner review for adults with asthma. Cochrane Database Syst Rev. 2003;(1):CD001117. doi: 10.1002/14651858.CD001117. PMID 12535399
- [Background] Ellis SE, Speroff T, Dittus RS, Brown A, Pichert JW, Elasy TA. Diabetes patient education: a meta-analysis and meta-regression. Patient Educ Couns. 2004 Jan;52(1):97-105. doi: 10.1016/s0738-3991(03)00016-8. PMID 14729296
- [Background] Gary TL, Genkinger JM, Guallar E, Peyrot M, Brancati FL. Meta-analysis of randomized educational and behavioral interventions in type 2 diabetes. Diabetes Educ. 2003 May-Jun;29(3):488-501. doi: 10.1177/014572170302900313. PMID 12854339
- [Background] Smith SM, Allwright S, O'Dowd T. Effectiveness of shared care across the interface between primary and specialty care in chronic disease management. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004910. doi: 10.1002/14651858.CD004910.pub2. PMID 17636778
- [Background] Oelke ND, Cunning L, Andrews K, Martin D, MacKay A, Kuschminder K, Congdon V. Organizing care across the continuum: primary care, specialty services, acute and long-term care. Healthc Q. 2009;13 Spec No:75-9. doi: 10.12927/hcq.2009.21102. PMID 20057254
- [Background] Delon S, Mackinnon B; Alberta Health CDM Advisory Committee. Alberta's systems approach to chronic disease management and prevention utilizing the expanded chronic care model. Healthc Q. 2009;13 Spec No:98-104. doi: 10.12927/hcq.2009.21106. PMID 20057258
- [Background] Walsh K, Duke J, Foureur M, Macdonald L. Designing an effective evaluation plan: a tool for understanding and planning evaluations for complex nursing contexts. Contemp Nurse. 2007 May-Jun;25(1-2):136-45. doi: 10.5172/conu.2007.25.1-2.136. PMID 17622997
- [Background] Nolte S, Elsworth GR, Sinclair AJ, Osborne RH. The extent and breadth of benefits from participating in chronic disease self-management courses: a national patient-reported outcomes survey. Patient Educ Couns. 2007 Mar;65(3):351-60. doi: 10.1016/j.pec.2006.08.016. Epub 2006 Oct 5. PMID 17027221
- [Derived] Contant E, Loignon C, Bouhali T, Almirall J, Fortin M. A multidisciplinary self-management intervention among patients with multimorbidity and the impact of socioeconomic factors on results. BMC Fam Pract. 2019 Apr 22;20(1):53. doi: 10.1186/s12875-019-0943-6. PMID 31010425
- [Derived] Fortin M, Chouinard MC, Diallo BB, Bouhali T. Integration of chronic disease prevention and management services into primary care (PR1MaC): findings from an embedded qualitative study. BMC Fam Pract. 2019 Jan 9;20(1):7. doi: 10.1186/s12875-018-0898-z. PMID 30626313
- [Derived] Fortin M, Chouinard MC, Dubois MF, Belanger M, Almirall J, Bouhali T, Sasseville M. Integration of chronic disease prevention and management services into primary care: a pragmatic randomized controlled trial (PR1MaC). CMAJ Open. 2016 Oct 12;4(4):E588-E598. doi: 10.9778/cmajo.20160031. eCollection 2016 Oct-Dec. PMID 28018871
- [Derived] Fortin M, Chouinard MC, Bouhali T, Dubois MF, Gagnon C, Belanger M. Evaluating the integration of chronic disease prevention and management services into primary health care. BMC Health Serv Res. 2013 Apr 8;13:132. doi: 10.1186/1472-6963-13-132. PMID 23565674
- See also: CIHR Applied Research Chair - Health Services and Policy Research on Chronic Diseases in Primary Care — http://www.usherbrooke.ca/crmcspl/en/
- See also: Agence de la santé et des services sociaux du Saguenay-Lac-Saint-Jean — http://www.santesaglac.gouv.qc.ca/
- See also: Université de Sherbrooke — http://www.usherbrooke.ca
- See also: Université du Québec à Chicoutimi — http://www.uqac.ca